CLINICAL TRIAL: NCT03558295
Title: CHoosing Triple or Double therApy in the Era of nOac for patientS Undergoing PCI: the CHAOS a Multicenter Study.
Brief Title: CHAOS Registry Study
Acronym: CHAOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Principal Investigator, A.O.U. Città della Salute e della Scienza
Other Study IDs: CHAOS
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Ischem Heart Disease; Primary Coronay Intervention; Oral Anticoagulants; Atrial Fibrillation
Keywords: Percutaneous coronary intervention (PCI), oral anticoagulants, atrial fibrillation, DOAC.
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Oral Anticoagulant — warfarin, dabigatran, rivaroxaban, edoxaban

SUMMARY:
INTRODUCTION: About 6-8% of patients undergoing PCI have an indication for long-term oral anticoagulants (OACs) due to various conditions such as atrial fibrillation (AF), mechanical heart valves, or venous thromboembolism. The addition of single or double antiplatelet therapy to OACs therapy results in an increase in bleeding complications (1-4). The standard of care of management in this patients, indicated by 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease (5), recommends the use of a triple therapy (Aspirin, clopidogrel and OAC) for 1-6 months (depending on the ischemic and hemorrhagic risk), then continue with double therapy only up to twelve month (Aspirin or clopidogrel and OAC) and after twelve months continue with the OAC only; the use of prasugrel or ticagrelor as part of triple therapy should be avoided (6). Only RELY study enrolled a small number of patients, less than one thousand, treated with dabigatran plus DAPT. Moreover, In the recent RCTs (WOEST(7), PIONEER AF-PCI study(8) and REDUAL-PCI(9)) only the double therapy (Aspirin or Clopidogrel/ticagrelor and DOAC) against triple therapy with warfarin was tested; and furthermore patients enrolled in RCTs represent only a small and not always representative sample of people treated in everyday clinical practice, who report a large burden of comorbidities and an older age. Randomized head to head comparison of warfarin and DOACs life-long (over 12 months from the PCI) have not been performed yet with clinical events as end points.

AIMS: Aim of the present study is to describe the contemporary management of patients who underwent a PCI and have an indication to OAC for AF evaluating the different types of combination therapies used (triple therapy with warfarin or with DOAC, single anti-platelet therapy plus warfarin or DOAC) and their management in the first year after a PCI in a "real-life" setting. Secondary we would also evaluate the safety (in term of bleedings) and the efficacy (in term of ischemic and cardioembolic events) of the use of the different combination of single or double antiplatelet with OACs, in patients with coronary artery disease.

MATERIALS AND METHODS: This is a retrospective, multicenter study including patients presenting with coronary artery disease (acute or stable setting) undergoing to PCI, in single or double antiplatelet therapy (aspirin, clopidogrel, ticagrelor, prasugrel, aspirin and clopidogrel, aspirin and ticagrelor, aspirin and prasugrel) with an indication to anticoagulant therapy (warfarin, dabigatran, rivaroxaban, edoxaban). The different groups will be compared with a propensity score analysis with matching.

Primary (efficacy) end-points:

* A composite end points including death, myocardial infarction, stent thrombosis, revascularization stroke (MACE).
* A composite end points including death, myocardial infarction, stent thrombosis, revascularization, stroke and BARC [Bleedings according to the Bleeding Academic Research Consortium] 2,3,5 (7,8): all events mutually exclusive (NACE).

Secondary end-points: Individual components of NACE; Cardiac death; Stroke; Target vessel revascularization (TVR) and non TVR and the number of the revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with final diagnosis of CAD (stable CAD or ACS) treated with oral anticoagulants and who undwerwent a coronary artery intervention
* Age ≥ 18 years
* Obtained informed consent

Exclusion Criteria:

* Oral anticoagulation indication other than atrial fibrillation
* Patients who underwent revascularization with thrombolysis or with BPAC
* Patients in active treatment with anti-cancer therapy
* Patients with a non obstructive coronary artery disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease (acute or stable setting) in single or double antiplatelet therapy (aspirin, clopidogrel, ticagrelor, prasugrel, aspirin and clopidogrel, aspirin and ticagrelor, aspirin and prasugrel) associated with oral anticoagulant (warfarin, dabigatran, rivaroxaban, edoxaban)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary (efficacy and safety) end-points:Net Adverse Clinical Event - NACE | 12 months
  Primary (efficacy and safety) end-points:
  - Net Adverse Clinical Event - NACE at 12 months of follow up (a composite end points including death, myocardial infarction, stent thrombosis, revascularization, stroke and BARC [Bleedings according to the Bleeding Academic Research Consortium] 2,3,5 (8,9): all events mutually exclusive); expressed as a rate of events.
Primary (efficacy and safety) end-points:Major Adverse Cardiac Event - MACE at 12 months | 12 months
  Primary (efficacy and safety) end-points:
  - Major Adverse Cardiac Event - MACE at 12 months of follow up (a composite end points including death, myocardial infarction (excluding periprocedural myocardial infarction), stent thrombosis, revascularization, stroke); expressed as a rate of events.

SECONDARY OUTCOMES:
Cardiac death | after 12 months
  Expressed as a rate of events.
Target vessel revascularization (TVR) and non TVR and the number of the revascularization. | after 12 months
  Expressed as a rate of events.
Death | after 12 months
  Expressed as a rate of events.
Myocardial infarction | after 12 months
  Expressed as a rate of events.
Stent thrombosis | after 12 months
  Expressed as a rate of events.
Recurrent revascularization | after 12 months
  Expressed as a rate of events.
Stroke | after 12 months
  Expressed as a rate of events.
Bleeding BARC [Bleedings according to the Bleeding Academic Research Consortium] 2,3,5 (8,9): all events mutually exclusive); expressed as a rate of events. | after 12 months
  According with BARC [Bleedings according to the Bleeding Academic Research Consortium] 2,3,5 (8,9): all events mutually exclusive); expressed as a rate of events.

CONTACTS AND LOCATIONS:
Locations (1):
- Città della Salute e della Scienza di Torino, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sorensen R, Hansen ML, Abildstrom SZ, Hvelplund A, Andersson C, Jorgensen C, Madsen JK, Hansen PR, Kober L, Torp-Pedersen C, Gislason GH. Risk of bleeding in patients with acute myocardial infarction treated with different combinations of aspirin, clopidogrel, and vitamin K antagonists in Denmark: a retrospective analysis of nationwide registry data. Lancet. 2009 Dec 12;374(9706):1967-74. doi: 10.1016/S0140-6736(09)61751-7. PMID 20006130
- [Result] Hansen ML, Sorensen R, Clausen MT, Fog-Petersen ML, Raunso J, Gadsboll N, Gislason GH, Folke F, Andersen SS, Schramm TK, Abildstrom SZ, Poulsen HE, Kober L, Torp-Pedersen C. Risk of bleeding with single, dual, or triple therapy with warfarin, aspirin, and clopidogrel in patients with atrial fibrillation. Arch Intern Med. 2010 Sep 13;170(16):1433-41. doi: 10.1001/archinternmed.2010.271. PMID 20837828
- [Result] Dans AL, Connolly SJ, Wallentin L, Yang S, Nakamya J, Brueckmann M, Ezekowitz M, Oldgren J, Eikelboom JW, Reilly PA, Yusuf S. Concomitant use of antiplatelet therapy with dabigatran or warfarin in the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) trial. Circulation. 2013 Feb 5;127(5):634-40. doi: 10.1161/CIRCULATIONAHA.112.115386. Epub 2012 Dec 27. PMID 23271794
- [Result] Oldgren J, Budaj A, Granger CB, Khder Y, Roberts J, Siegbahn A, Tijssen JG, Van de Werf F, Wallentin L; RE-DEEM Investigators. Dabigatran vs. placebo in patients with acute coronary syndromes on dual antiplatelet therapy: a randomized, double-blind, phase II trial. Eur Heart J. 2011 Nov;32(22):2781-9. doi: 10.1093/eurheartj/ehr113. Epub 2011 May 7. PMID 21551462
- [Result] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):34-78. doi: 10.1093/ejcts/ezx334. No abstract available. PMID 29045581
- [Result] Sarafoff N, Martischnig A, Wealer J, Mayer K, Mehilli J, Sibbing D, Kastrati A. Triple therapy with aspirin, prasugrel, and vitamin K antagonists in patients with drug-eluting stent implantation and an indication for oral anticoagulation. J Am Coll Cardiol. 2013 May 21;61(20):2060-6. doi: 10.1016/j.jacc.2013.02.036. Epub 2013 Mar 21. PMID 23524219
- [Result] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Result] Dewilde WJ, Oirbans T, Verheugt FW, Kelder JC, De Smet BJ, Herrman JP, Adriaenssens T, Vrolix M, Heestermans AA, Vis MM, Tijsen JG, van 't Hof AW, ten Berg JM; WOEST study investigators. Use of clopidogrel with or without aspirin in patients taking oral anticoagulant therapy and undergoing percutaneous coronary intervention: an open-label, randomised, controlled trial. Lancet. 2013 Mar 30;381(9872):1107-15. doi: 10.1016/S0140-6736(12)62177-1. Epub 2013 Feb 13. PMID 23415013
- [Result] Gibson CM, Mehran R, Bode C, Halperin J, Verheugt FW, Wildgoose P, Birmingham M, Ianus J, Burton P, van Eickels M, Korjian S, Daaboul Y, Lip GY, Cohen M, Husted S, Peterson ED, Fox KA. Prevention of Bleeding in Patients with Atrial Fibrillation Undergoing PCI. N Engl J Med. 2016 Dec 22;375(25):2423-2434. doi: 10.1056/NEJMoa1611594. Epub 2016 Nov 14. PMID 27959713
- [Result] Cannon CP, Bhatt DL, Oldgren J, Lip GYH, Ellis SG, Kimura T, Maeng M, Merkely B, Zeymer U, Gropper S, Nordaby M, Kleine E, Harper R, Manassie J, Januzzi JL, Ten Berg JM, Steg PG, Hohnloser SH; RE-DUAL PCI Steering Committee and Investigators. Dual Antithrombotic Therapy with Dabigatran after PCI in Atrial Fibrillation. N Engl J Med. 2017 Oct 19;377(16):1513-1524. doi: 10.1056/NEJMoa1708454. Epub 2017 Aug 27. PMID 28844193
- [Result] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487